CLINICAL TRIAL: NCT06922422
Title: The Effects of Sensory-Motor Integration Exercises on Sensory Processing and Balance in Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Sensory-Motor Integration for Sensory Processing and Balance in ASD
Acronym: SMIE-ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: King Saud University (Other); Taif University (Other)
Responsible Party: Principal Investigator, Mohamed Aly, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EgyCTR102024002
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Interventions:
  * Experimental: Sensory-Motor Integration Exercises
  * Sessions: 64 (45 min/session, 4 days/week)
  * Duration: 16 weeks
  * Components: Tactile, proprioceptive, and vestibular activities designed for individual sensory profiles.
  * Active Comparator: Conventional Therapy
  * Applied Behavior Analysis (ABA)
  * Massage therapy
  * Sessions: Same duration (45 min/session, 4 days/week)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants received structured sensory-motor integration exercises, consisting of sensory play activities tailored to enhance sensory processing and balance. Sessions lasted 45 minutes each, conducted 4 times weekly for 16 weeks (64 total sessions).
  Interventions: Behavioral: Sensory-Motor Integration Exercises
- Control group (Active Comparator): Participants received conventional therapy including Applied Behavior Analysis (ABA) and massage therapy, conducted for 45 minutes per session, 4 times weekly, for 16 weeks (64 total sessions). These sessions did not include sensory-specific interventions.
  Interventions: Behavioral: Conventional therapy group

INTERVENTIONS:
Behavioral: Sensory-Motor Integration Exercises — A structured sensory-motor integration program based on sensory play activities designed to enhance sensory processing and balance. Each session lasted 45 minutes, conducted four times per week, for a total of 64 sessions over 16 weeks. Activities targeted multiple sensory modalities, including tactile, proprioceptive, and vestibular inputs.
  Arms: Intervention group
Behavioral: Conventional therapy group — Conventional therapy sessions consisting of Applied Behavior Analysis (ABA) and massage therapy without specific sensory-motor integration activities. Each session lasted 45 minutes, conducted four times weekly, for a total of 64 sessions over 16 weeks.
  Arms: Control group

SUMMARY:
This randomized controlled trial evaluates the effectiveness of a 16-week structured sensory-motor integration exercise program compared to conventional therapy (Applied Behavior Analysis and massage therapy) in improving sensory processing abilities and balance in children aged 6-12 years diagnosed with Autism Spectrum Disorder (ASD). Outcomes are measured using the Short Sensory Profile and Berg Balance Scale at baseline and after 16 weeks of intervention. Findings aim to demonstrate the clinical utility of sensory-motor integration exercises in enhancing functional outcomes for children with ASD.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder often experience significant sensory processing issues and motor coordination challenges, particularly balance deficits. This study evaluates a sensory-motor integration intervention aimed at improving sensory modulation and motor abilities. Participants aged 6 to 12 years are randomized into two groups: an intervention group participating in structured sensory-motor exercises (64 sessions, 4 times weekly, 45 minutes per session), and a control group receiving conventional therapy (primarily Applied Behavior Analysis and massage therapy). Outcomes are assessed using standardized measures: the Short Sensory Profile (SSP) for sensory processing and the Berg Balance Scale (BBS) for balance, at baseline and immediately following the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years
* Diagnosed with Autism Spectrum Disorder (DSM-5 criteria)
* Mild-to-moderate ASD severity (CARS score ≤ 39.5)
* Ability to participate in structured sessions

Exclusion Criteria:

* Significant physical impairments or medical conditions affecting participation
* Recent (within 6 months) participation in sensory integration therapy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Short Sensory Profile (SSP) | 16 weeks
  Change in sensory processing
Berg Balance Scale (BBS) | 16 weeks
  Change in functional balance

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Sciences, Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected during the trial will be shared, including baseline characteristics, Short Sensory Profile (SSP) scores, and Berg Balance Scale (BBS) outcomes. No personally identifiable information will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting documents will be made available beginning 6 months after publication of the primary results and will remain accessible for at least 5 years.
Access Criteria: Qualified researchers and healthcare professionals can request access to the data for scientific purposes. Requests should include a brief research proposal and data use agreement. Access will be granted through a secure platform or upon direct request to the principal investigator.